CLINICAL TRIAL: NCT05537142
Title: A Phase I, Open-label, Single-center, Single-dose, Parallel Group Study to Evaluate the Pharmacokinetics of BV100 in Participants with Mild, Moderate, and Severe Hepatic Impairment Compared to Matched Healthy Control Participants
Brief Title: A Study to Assess the Phamacokinetics of BV100 in Participants with Varying Degrees of Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioVersys AG (Industry)
Collaborators: Clinical Research Units Hungary (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BV100-008
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-05

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Experimental): Participants with Normal hepatic Function
  Interventions: Drug: BV100
- Group 2 (Experimental): Participants with mild hepatic impairment: Child-Pugh A (Score 5-6)
  Interventions: Drug: BV100
- Group 3 (Experimental): Participants with moderate hepatic impairment: Child-Pugh B (Score 7-9)
  Interventions: Drug: BV100
- Group 4 (Experimental): Participants with severe hepatic impairment: Child-Pugh C (Score 10-15)
  Interventions: Drug: BV100

INTERVENTIONS:
Drug: BV100 — Rifabutin for Infusion

SUMMARY:
To investigate the pharmacokinetics (PK) of rifabutin in subjects with hepatic impairment after single intravenous (IV) infusion of BV100

DETAILED DESCRIPTION:
To investigate the pharmacokinetics (PK) of rifabutin and excipient in subjects with hepatic impairment after single intravenous (IV) infusion of BV100. In addition to investigate the safety and tolerability of BV100 in subjects with hepatic impairment and to investigate the PK of 25-deacetyl-rifabutin metabolite in subjects with hepatic impairment after single intravenous (IV) infusion of BV100

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria will be:

All participants (Groups 1-4):

1. Participants must provide written informed consent prior to any screening procedures being performed.
2. Male and non-child bearing potential females between 18 and 75 years of age, inclusive
3. Women of non-childbearing potential is defined as women who are physiologically and/or anatomically incapable of becoming pregnant, as now further described:

   * They are post-menopausal as evidenced by 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate history of vasomotor symptoms).
   * They have had bilateral surgical oophorectomy (with or without hysterectomy), total hysterectomy or bilateral tubal ligation at least six weeks prior. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment she is considered not of childbearing potential.
4. Participants must weigh at least 50.0 kg and must have a BMI within the range of 18.0 to 38.0 kg/m2, inclusive, for healthy participants at Screening. For hepatic impairment participants without overt ascites, the BMI should be within the range of 18 to 40 kg/m2. For hepatic impairment participants with overt ascites, the BMI should be within the range of 18 to 45 kg/m2
5. Participant is able to read, speak, and understand the local language, to understand and comply with the requirements of the study.
6. Must be a non-smoker or agree to smoke no more than 10 cigarettes or equivalent nicotine containing products per day and are committed not to increase the consumption during the study period

   Additional inclusion criteria for healthy participants (Group 1):
7. Each participant must match in age (+/- 10 years), gender, weight (+/- 20%), and smoking status to a participant in Groups 2, 3 and/or 4.
8. Seated vital signs must be within the following ranges at Screening and Baseline:

   * Body temperature, 35.0 to 37.5°C, inclusive
   * Systolic blood pressure, 89 to 140 mmHg, inclusive
   * Diastolic blood pressure, 50 to 90 mmHg, inclusive
   * Pulse rate, 40 to 100 bpm, inclusive
9. Healthy participants with no clinically significant abnormalities as determined by past medical history, physical examination, vital signs, ECG, and clinical laboratory test

   Additional inclusion criteria for mild, moderate and severe hepatic impairment participants (Groups 2-4):
10. Participants with Child-Pugh Clinical Assessment Score as calculated per the Child-Pugh classification.
11. Seated vital signs must be within the following ranges at Screening and Baseline:

    * Body temperature, 35.0 to 37.5°C, inclusive
    * Systolic blood pressure, 89 to 160 mmHg, inclusive
    * Diastolic blood pressure, 50 to 100 mmHg, inclusive
    * Pulse rate, 40 to 100 bpm, inclusive
12. Stable Child-Pugh status at Screening and Baseline visits
13. Participants with impaired hepatic function and other stable medical disorders such as diabetes, hypertension, hyperlipidemia, hypothyroidism etc., are eligible, as long as they are considered appropriate for enrollment, as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at Screening and Baseline

Exclusion Criteria:

The main exclusion criteria will be:

All participants (Groups 1-4):

1. Contraindication or hypersensitivity to the investigational compound/compound class or excipients being used in this study.
2. Woman of childbearing potential, or pregnant or lactating females.
3. Sexually active males unless they use a condom during intercourse for 8 weeks after BV100 intake and must not father a child in this 8 week period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid. In addition, male participants must not donate sperm for 8 weeks after study drug intake.
4. History or presence of clinically significant ECG abnormalities or a family history or presence of prolonged QT-interval syndrome.
5. Abnormal ECG findings at Screening:

   * Clinically significant ST/T wave abnormalities as determined by the Investigator
   * Inability to determine the QT interval on ECG
   * Specific to hepatic impaired patients:

     o QTcF > 480 ms (males and females)
   * Specific to healthy control participants:

     * PR > 220 ms, QRS complex > 120 ms, QTcF > 450ms for males; QTcF > 470ms for females.
6. Clinically significant cardiac conduction abnormality as determined by the Investigator
7. History of clinically significant cardiovascular disease (e.g., congestive heart failure NYHA Class II-IV, atherosclerosis, labile hypertension or uncontrolled hypertension)
8. History of psychiatric illness within the past 2 years that may interfere with the ability to comply with the protocol requirements.
9. History of malignancy of any organ system, treated or untreated, within 3 years, regardless of whether there is recurrence or metastases. Those with localized basal cell carcinoma of the skin, in-situ cervical cancer, or hepatocellular cancer treated with local ablative therapy more than 6 months ago may be enrolled.
10. Recent (within the last 3 years of Screening) or recurrent history of autonomic dysfunction (e.g. recurrent episodes of fainting palpitations).
11. History of immunodeficiency diseases, including a positive HIV test result.
12. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardize the participant in case of participation in the study.
13. History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, bowel resection or cholecystectomy (cholecystectomy allowed for severe participants only)
14. History of, or clinical evidence of, pancreatic injury or pancreatitis within the preceding 1 month prior to dosing
15. Evidence of urinary obstruction or difficulty in voiding at screening
16. Use of investigational drugs (i.e., participation in any clinical investigation) within 4 weeks prior to dosing or longer if required by local regulation, or within 5 half-lives of the investigational agent taken prior to dosing (whichever is longer).
17. Consumption of Seville oranges, grapefruit, grapefruit juices, grapefruit hybrids, pomelos, pomegranates, star fruit, or exotic fruits (as well as their juices) and cruciferous vegetables (such as Brussel sprouts, broccoli, cabbage, cauliflower) for 14 days prior to dosing until completion of the End of Study Visit. The juices (except for orange juice) and products containing these fruits must also be avoided.
18. Administration of medications that prolong the QT interval within 14 days or 5 half-lives, whichever is longer, prior to dosing and throughout the study.
19. Use of any live vaccines against infectious diseases within 4 weeks of initiation of study treatment. Coronavirus disease (COVID-19) vaccines will be restricted within 2 weeks prior to dosing of study treatment until completion of the End of Study visit.
20. Participants not willing to abstain from alcohol 48 hours prior to dosing, confirmed by alcohol breath test at baseline, and until after Study Completion evaluation.
21. Participants with known ongoing alcohol and/or drug abuse within 1 month prior to Screening or evidence of such abuse as indicated by the laboratory assays conducted during the screening or baseline evaluations. For participants with impaired hepatic function (groups 2-4), participation in the study may be allowed, if the positive drug screen is due to prescription drug use for a specific symptom such as insomnia or pain. Unhealthy alcohol use is defined as use more than 24g pure alcohol per day for male and 12 g for female (12 g equals to approximately 300 mL beer, 100 mL wine, or 25 mL spirits).
22. Donation or loss of 500 mL or more of blood within 8 weeks prior to dosing.
23. Potentially unreliable or vulnerable participants (e.g., person kept in detention) and those judged by the investigator to be unsuitable for the study.
24. Participant has positive Coronavirus (SARS-CoV-2) rapid test and positive PCR test upon Check-in on Day-1.
25. Participant who had severe course of COVID-19 (e.g., hospitalisation and/or extra-corporeal membrane oxygenation, mechanically ventilated) within 2 months prior to Screening.
26. Acute hepatitis B or C infection at Screening or active infection requiring therapy that will not be completed before screening.

    Additional exclusion criteria for healthy participants (Group 1):
27. Significant illness within the 2 weeks prior to dosing
28. ALT, AST, GGT, or ALP ≥ 1.2 ULN OR total bilirubin ≥ ULN OR any elevation ≥ ULN of more than one parameter among ALT, AST, GGT or ALP at Screening or Baseline.
29. Participants known to have Gilbert´s syndrome.
30. Hemoglobin levels below ≤ LLN at Screening or Baseline (unless deemed not clinically significant by the investigator).
31. Platelet count ≤ LLN at Screening or Baseline (unless deemed not clinically significant by the investigator).
32. Presence of impaired renal function as indicated by serum creatinine > ULN or abnormal urinary constituents (e.g., albuminuria) at Screening.
33. Chronic hepatitis B or hepatitis C infection.
34. Intake of any prescription or non-prescription medication, dietary supplements, vitamins or herbal remedies within 2 weeks prior to the dosing of study treatment and within 4 weeks prior to dosing for treatment known to affect CYP3A4. Limited use of acetaminophen (up to 2g/day) is acceptable but must be documented in the Concomitant Medications/Significant non-drug therapies page of the electronic Case Report Forms (eCRF).

    Mild and moderate hepatic impairment participants (Groups 2-3):
35. Participants with hepatic impairment with abnormal laboratory values for the following parameters at Screening or Baseline:

    * Hemoglobin < 9 g/dL.
    * Platelet count < 30 × 109/L.
    * White blood cell count < 2.5 × 109/L.
    * Total bilirubin > 8 mg/dL.
    * Serum amylase > 5 × ULN with no abdominal symptoms (>2 x ULN with abdominal symptoms)
    * International standardized ratio (INR) > 2.5.
    * Corrected serum calcium < 8.6 or > 10.2 mg/dL.
36. Severe complications of liver disease within the preceding 3 months prior to dosing.
37. Hospitalisation due to liver disease within the preceding 1 month prior to dosing.
38. Participant has received liver transplant at any time in the past and is on immunosuppressant therapy.
39. Participants requiring paracentesis more than every 3 weeks for the management of ascites are excluded. Participants who are receiving diuretics to manage ascites can be enrolled and will be assigned the Child-Pugh score for the degree of ascites while on diuretic treatment. The diuretic dose must have been stable for 7 days prior to dosing.
40. Transjugular intrahepatic portosystemic shunt and/or have undergone portacaval shunting.
41. Clinically significant abnormal findings in physical examination, ECG, or laboratory evaluations, not consistent with known clinical disease.
42. Significant change or addition to routine medication (prescribed) within 1 month prior to dosing, except for changes to medication that require frequent dose adjustments, such as insulin, furosemide (Lasix), Aldactone or analgesia, which can be made within 14 days prior to dosing, as agreed between the investigator and BioVersys.
43. Active Grade 3 or 4 hepatic encephalopathy within 1 month prior to dosing.
44. Primary biliary cholangitis or biliary obstruction.
45. History of gastrointestinal bleeding requiring hospitalisation within the past 3 months prior to Screening.
46. Presence of moderate to severe impaired renal function as indicated by any or all of the following criteria:

    * Creatinine clearance < 50 mL/min as calculated using the Cockcroft-Gault formula or eGFR < 50 mL/min/1.73 m2 based on CK-EPI calculation.
    * Serum creatinine > 1.5 × ULN.
47. Clinically significant abnormal findings in physical examination, ECG or laboratory evaluations, not consistent with known clinical disease
48. Clinically significant illness within 2 weeks prior to dosing that may jeopardize safety of the study participant and/or alter the study results as judged by the investigator
49. Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled di-abetes, active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with protocol
50. Participants with hepatic impairment may continue to receive medications required to treat their current disease upon confirmation by BioVersys, with exception of moderate or strong CYP3A4 inducers or inhibitors within 4 weeks prior to dosing until completion of the End of Study Visit.

    Severe hepatic impairment participants (Group 4):
51. Participants with hepatic impairment with abnormal laboratory values for the following parameters at Screening or Baseline:

    * Hemoglobin < 8.5 g/dL.
    * Platelet count < 30 × 109/L.
    * White blood cell count < 2.5 × 109/L.
    * Total bilirubin > 8 mg/dL.
    * Serum amylase > 5 × ULN with no abdominal symptoms (>2 x ULN with ab-dominal symptoms).
    * International standardized ratio (INR) > 2.5.
52. Severe complications of liver disease within the preceding 1 months prior to dosing.
53. Participant has received liver transplant at any time in the past and is on immunosuppressant therapy.
54. Participants requiring paracentesis more than every 3 weeks for the management of ascites are excluded. Participants who are receiving diuretics to manage ascites can be enrolled and will be assigned the Child-Pugh score for the degree of ascites while on diuretic treatment. The diuretic dose must have been stable for 7 days prior to dosing.
55. Transjugular intrahepatic portosystemic shunt and/or have undergone portacaval shunting.
56. Clinically significant abnormal findings in physical examination, ECG, or laboratory evaluations, not consistent with known clinical disease.
57. Significant change or addition to routine medication (prescribed) within 1 month prior to dosing, except for changes to medication that require frequent dose adjustments, such as insulin, furosemide (Lasix), Aldactone or analgesia, which can be made within 14 days prior to dosing, as agreed between the investigator and BioVersys.
58. Presence of moderate to severe impaired renal function as indicated by any or all of the following criteria:

    * Creatinine clearance < 50 mL/min as calculated using the Cockcroft-Gault formula or eGFR < 50 mL/min/1.73 m2 based on CK-EPI calculation.
    * Serum creatinine > 1.5 × ULN.
59. Active Grade 3 or 4 hepatic encephalopathy within 1 month prior to dosing.
60. Primary biliary cholangitis or biliary obstruction.
61. History of gastrointestinal bleeding requiring hospitalisation within the past 3 months prior to Screening.
62. Clinically significant illness within 2 weeks prior to dosing that may jeopardize safety of the study participant and/or alter the study results as judged by the investigator
63. Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled di-abetes, active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with protocol.
64. Participants with hepatic impairment may continue to receive medications required to treat their current disease upon confirmation by BioVersys, with exception of moderate or strong CYP3A4 inducers or inhibitors within 4 weeks prior to dosing until completion of the End of Study Visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
To investigate the pharmacokinetics (PK) of rifabutin in participants with hepatic impairment | 15 days
  Area under the plasma concentration versus time curve (AUC)
To characterize the single dose pharmacokinetic profile of rifabutin | 15 days
  Peak Plasma Concentration (Cmax)

SECONDARY OUTCOMES:
To investigate the safety and tolerability of single intravenous ascending doses of BV100 assessed by the nature, occurrence, and severity of treatment-emergent adverse events | 31 Days
  Safety and Tolerability
To determine the plasma concentration of the main metabolite 25-O-Desacetyl-Rifabutin in plasma in participants with hepatic impairment | 15 days
  Pharmacokinetics
To determine the plasma concentration of DMI in plasma in subjects with hepatic impairment | 15 days
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Geza Lakner, MD, Principal Investigator — Clinical Research Units Hungary
Locations (1):
- CRU Hungary Kft., Early Phase Unit, Kistarcsa, Hungary

IPD SHARING:
Plan to Share IPD: Undecided